CLINICAL TRIAL: NCT06437691
Title: Effect of Stent Placement on Short Term Survival of Left Sided Obstructive Colorectal Cancers. Comparison of Bridge-To-Surgery Versus Emergency Surgery Approaches
Brief Title: Effect of Stent Placement on Short Term Survival of Left Sided Obstructive Colorectal Cancers
Status: Completed | Type: Observational
Sponsor: Yasir Musa Kesgin, MD (Other)
Responsible Party: Sponsor-Investigator, Yasir Musa Kesgin, MD, MD, Kanuni Sultan Suleyman Training and Research Hospital
Organization: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Other Study IDs: StentSurv
Record Dates: First submitted 2024-05-25; First posted 2024-05-31 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Colorectal Cancer
Keywords: Obstruction, Bridge To Surgery
MeSH Terms: conditions — Colorectal Neoplasms; Bites and Stings

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A - Emergency Surgery Group: Patients underwent emergency surgery directly after coming to emergency department due to left sided obstructive colorectal cancer
- Group B - Stent Group: Left sided obstructive colorectal cancer patients underwent elective surgery following decompression via self-expandable metallic stent placement.
  Interventions: Procedure: Self-Expandable Metallic Stent Placement

INTERVENTIONS:
Procedure: Self-Expandable Metallic Stent Placement
  Groups: Group B - Stent Group

SUMMARY:
The aim of this observational study is to determine effect of stent placement on survival results in first three years in a patient who applied to the emergency department with obstruction due to colorectal cancer. Eligible patients divided into two groups. Group A includes patients underwent emergency surgery directly. Patients underwent elective surgery following stent placement as bridge-to-surgery. Patients underwent elective surgery following bridge-to-surgery stent placement were accepted as Group B.

DETAILED DESCRIPTION:
Patients who applied to emergency department of a single tertiary referral center between January 2016 and December 2020 and diagnosed as left sided obstructive colorectal cancer were included in this retrospective study. All patients were equal or older than 18 years and histopathologically found to have primary colorectal malignant neoplasms.

Patients were excluded from the analysis if they met any of the following criteria:

* Who underwent emergency surgery due to unsuccessful stent application intervention or stent-related complications developed,
* Those with middle and lower rectum tumors or received neoadjuvant treatment,
* Perforation,
* Who underwent subtotal or total colectomy (as a result of colon ischemia in the cecum, microperforation, etc.),
* Recurrent disease patients
* Patients have metastasis

ELIGIBILITY:
Inclusion Criteria:

* All patients were equal or older than 18 years and histopathologically found to have primary colorectal malignant neoplasms and diagnosed as left sided (descending colon, sigmoid colon and upper rectum) obstructive colorectal cancer were included

Exclusion Criteria:

* Who underwent emergency surgery due to unsuccessful stent placement intervention
* Who underwent emergency surgery due to stent-related complications
* Those with middle and lower rectum tumors
* Those received neoadjuvant treatment,
* Patients have perforation,
* Who underwent subtotal or total colectomy (as a result of colon ischemia in the cecum, microperforation, etc.),
* Who has a recurrent disease or metastasis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients come to emergency department and diagnosed as left sided obstructive colorectal cancer
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 3 years
  The survival time of patient after being diagnosed as colorectal cancer after coming to emergency department
Disease Free Survival | 3 years
  The local or systemic recurrence free time period of patient after being diagnosed as colorectal cancer after coming to emergency department

SECONDARY OUTCOMES:
Mortality | 90 days
  Death of patient in postoperative first three months
Serious complications | 90 days
  Postoperative complications of patients that have a Clavien-Dindo Score greater than or equal to 3
Minimally invasive surgery | 90 days
  Patients that found a chance for fully minimally invasive surgery for resection of colorectal cancer
End colostomy rate | 90 days
  Patients that have a end colostomy at the end of surgical resection of colorectal cancer

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Sürek, Study Chair — Bakırköy Dr. Sadi Konuk Training and Research Hospital

IPD SHARING:
Plan to Share IPD: No
The datasets generated and analysed during the current study are not publicly available due to institutional policies but are available from the contact person on reasonable request.